CLINICAL TRIAL: NCT00079521
Title: The Effect of Therapeutic Touch on Bone Formation in Postmenopausal Women After Wrist Fracture
Brief Title: Therapeutic Touch for Wrist Fractures in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P20AT000756-01P1 (NIH)
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2006-08

CONDITIONS: Osteoporosis; Fractures
Keywords: Bone Metabolism; Therapeutic Touch
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Therapeutic Touch

INTERVENTIONS:
Procedure: Therapeutic Touch

SUMMARY:
This study will evaluate the effectiveness of therapeutic touch in treating wrist fractures in women past menopause.

DETAILED DESCRIPTION:
In the United States, the use of complementary and alternative medicine (CAM) increased by approximately 25% between 1990 and 1997. The number of visits to CAM practitioners exceeded visits to primary care physicians by about 250 million in 1997. Energy medicine modalities, including therapeutic touch, healing touch, and reiki, are commonly utilized for conditions ranging from headache to cancer, yet understanding of the human energy field and how it may be used in healing is limited. This study will examine the effect of therapeutic touch on fracture healing in postmenopausal women.

Women will be enrolled in the study within one week of a wrist fracture and will receive either therapeutic touch or a sham (placebo) treatment daily for 3 weeks. Assessments will include blood and urine analysis and measures of pain and function in the affected wrist.

ELIGIBILITY:
Inclusion Criertia:

* Postmenopausal
* Wrist fracture within 1 week of study entry
* Able to travel to research center for daily treatment

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2003-03; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Karen M. Prestwood, MD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States